CLINICAL TRIAL: NCT04607499
Title: Pregnancy Registry in West China: a Hospital-based Database Linking Electronic Medical Records
Brief Title: Pregnancy Registry in West China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: West China Hospital (Other)
Collaborators: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Jing Tan, Associate professor of Chinese Evidence-based Medicine Center, West China Hospital
Other Study IDs: PRWC
Record Dates: First submitted 2020-10-24; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Pregnant Women
Keywords: Registry; Pregnant women; West China; Electronic medical records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women without intervention

SUMMARY:
With the Healthy China 2030 Plan for further reducing maternal mortality ratio (MMR), and increasing number of high-risk pregnancies in China, we aimed to develop a registry of pregnant women based on hospital-based Electronic Medical Records (EMR) data in West China, through integrating information technology and medical knowledge, by linking multi-resource data covering information regarding the whole cycle from pregnancy registration till delivery, and process of diagnosis, treatment and pregnancy outcomes, in order to provide reliable, valuable and efficient data resources for researches about high-risk pregnancy safety and MMR reduction in southwestern China.

From January 29, 2014 to November 29, 2019, 64,468 pregnancies of 62,690 women were registered around gestational 13th weeks in the hospital, collecting over 47 million records (including repeated measurement data) from Health Information System (HIS), Laboratory Information System (LIS), and Picture Archiving and Communication System (PACS). After excluding 3476 pregnancies lost to follow-up and 7325 newly-pregnancies with expected date of delivery out of the study time, a total of 53,667 pregnancies about 51,964 women were finally included in the registry, who had been followed up till the occurrence of at least one outcome, including any pregnancy complication, abortion, stillbirth, induced labor, and live birth between January 1, 2015 and November 30, 2019.

Till now, through data linkage, data collection, cleaning and recoding, we have generated more than 2100 structured variables regarding pre-pregnancy conditions, prenatal visit records, hospitalized diagnosis, treatment and discharge outcomes. The diagnoses of pregnancy complications, maternal and fetal outcomes, recorded by ICD-10 coding or free terms in original fields, were uniformly encoded by the Classification and Codes of Diseases released by Chinese National Standards Institute (GB/T14396-2016) and National Health Standard Criteria for Birth Defects (WS 377.6-2013).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who registered prenatal information during first trimester at target hospital, and had been followed up till the occurrence of at least one outcome, including any pregnancy complication, abortion, stillbirth, induced labor, and live birth.

Exclusion Criteria:

* They only registered in the hospital, but lost to follow-up for various reasons, such as transferring out for treatment or delivery; or they were hospitalized for termination of pregnancy (e.g. induced labor) or treatment of any complications (e.g. pregnancy-induced hypertension syndrome), but had no pregnancy registry records at the first trimester; or they registered pre-pregnancy information in the hospital just before the end of the study, none of pregnancy outcomes such as live-birth delivery, has been followed-up within the study period.

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant women who registered prenatal information during first trimester at the West China Second University Hospital of Sichuan University, and had been followed up till the occurrence of at least one outcome, including any pregnancy complication, abortion, stillbirth, induced labor, and live birth.
Sampling Method: Probability Sample
Enrollment: 53667 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of pre-eclampsia | 22 weeks
  Maternal systolic blood pressure ≥ 140 mmHg and (or) diastolic pressure ≥ 90 mmHg, accompanied by any one of the following: urinary protein ≥ 0.3g/24 h, or the ratio of urinary protein and creatinine ≥ 0.3, or random urine protein ≥ (+) if quantitative urine protein is not available; no proteinuria but with any damages of heart, lung, liver, kidney and other important organs, or with abnormal changes of blood system, digestive system and nervous system, or placenta fetus involvement, etc.
Incidence of eclampsia | 22 weeks
  Tonic-clonic seizures (convulsions) in preeclampsia patients, including convulsions and coma, not due to pre-existing or organic brain disorders.
Incidence of gestational diabetes | 20 weeks
  By oral glucose tolerance test between 24 and 28 gestational weeks (fasting glucose ≥5.1 mmol/L, 1-h glucose ≥10.0 mmol/L, 2-h glucose ≥8.5 mmol/L; one abnormal result sufficient).
Incidence of ruptured uterus | Up to 40 weeks
  Rupture of maternal uterus confirmed by laparotomy.
Incidence of postpartum hemorrhage | Within 24h after delivery
  Postpartum bleeding volume ≥500 mL.
Incidence of maternal death | Up to 40 weeks
  Maternal death
Incidence of birth defects | Up to 40 weeks
  Birth defects such as anencephaly, spina bifida, encephalocele, hydrocephalus, cleft palate, cleft lip, microtia, esophageal atresia or stenosis, anorectal, hypospadias, ectropion of bladder, talipes equinovarus, polydactylism, ankylodactylia, congenital diaphragmatic hernia, umbilical cord prolapse, gastroschisis, conjoined twins, down syndrome, congenital heart disease, or other birth defects.
Incidence of preterm birth | Up to 37 weeks
  Delivery before 37th gestational weeks.
Value of neonatal birth weight | Within 24h after delivery
  Neonatal birth weight measured after birth.
Incidence of neonatal death | Within 28 days after delivery
  Neonatal death
Incidence of stillbirth | Up to 40 weeks
  Fetus death at or after 20-28 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghui Liu, MD, Study Director — West China Second University Hospital

IPD SHARING:
Plan to Share IPD: Yes
Research institutions could apply for data access by submitting a formal study protocol, subjected to approval by the West China Second University Hospital of Sichuan University and the Chinese Evidence-based Medicine Center of West China Hospital. Ethical review and research registration are mandatory for all studies.
Time Frame: The data will be available after study completion.